CLINICAL TRIAL: NCT02617173
Title: The Effect of Low Electrical Current on Testicular Spermatocyte Count
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-15-2514-GR-CTIL
Record Dates: First submitted 2015-11-22; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Oligozoospermia; Azoospermia
MeSH Terms: conditions — Oligospermia; Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcutaneous electrical nerve stimulation (Experimental): Low current electrical stimulator
  Interventions: Device: Micro 400 Matrix Therapy Products

INTERVENTIONS:
Device: Micro 400 Matrix Therapy Products — Positive electrical current with a low amplitude bellow sensation level situated on the scrotum.

SUMMARY:
Oligozoospermia, refers to a low concentration of sperm. A low sperm count or poor sperm quality is the cause of infertility in about 20% of couples with fertility problems, and a contributory factor in a further 25% of couples. In the majority of cases, no cause can be found. For mild male infertility, intra uterine insemination (IUI) is the procedure of choice with a pregnancy rate of 6.5%. In IUI, sperm is inserted using a thin, flexible catheter directly into a woman's uterus.

Azoospermia affects 1% of the male population and 20% of male infertility situations. Over 50% of azoospermic cases are due to testicular failure, including absence or failed production as well as low production and maturation arrest during the process of spermatogenesis. ICSI allows successful fertilization even with immature sperm obtained directly from testicular tissue. This is done through TESA (Testicular sperm aspiration) or TESE (Testicular sperm extraction). In cases of TESE small strips of testicular tissue are extracted with the intention of finding few viable sperm cells to be used for IVF or ICSI. Men with non-obstructive azoospermia have 0 to 3 mature spermatids per seminiferous tubule in contrast to 17-35 mature spermatids in men with normal spermatogenesis. TESE success rates are approximately 50% but differ according to etiology. Unfortunately, there is no method of pointing out where sperm may be found. TESE is accompanied with pain, tissue loss, reduced success in future TESE due to tissue scaring and testosterone deficiency.

The complex process of spermatogenesis includes maturation of young spermatids into spermatozoas, a process which takes approximately 74 days. During spermatogenesis, spermatogonial stem cells are transformed into spermatids and released from the seminiferous tubule epithelium into its lumen. Non-motile spermatozoa are transported through the seminifreous tubules to the epididymis by testicular fluid secreted from the Sertoli cells with the aid of peristaltic contraction. During transport through the epididymis, sperm cells develop the ability to progress forward, undergo capacitation and attach and penetrate the egg.

The electric charge of the spermatic cell has been termed zeta potential (electrokinetic potential) and is defined as the electric potential in the slip plane between the sperm membrane and its surroundings. Mature sperm possess an electric charge of -16 to -20 mV.

In the animal study conducted, positive electrical current with a low amplitude bellow sensation level was situated around the scrotum of four normospermic and one oligospermic male pigs. At the end of the research the concentration of spermatocytes in the epididymis obtained in surgery was found to be 200 to 1600 percent above the baseline.

Our intention is to evaluate if positive electrical current with a low amplitude bellow sensation level situated on the scrotum will increase the concentration of spermatocytes in the ejaculate.

If our hypothesis is confirmed this may become a method for treating male infertility. The period of improvement is still unclear.

ELIGIBILITY:
Inclusion Criteria:

* Men with primary infertility defined as a state of Azoospermia.
* Men with pathological sperm tests indices as defined by the WHO.

Exclusion Criteria:

* Men with genetic syndromes, and states of Azoospermia secondary to chemotherapy, bone marrow transplantation or radiation.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Spermatomcyte count in the ejaculate. | One year.
  To evaluate if positive electrical current with a low amplitude below sensation level situated on the scrotum will increase the concentration of spermatocytes in the ejaculate.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Raviv, Prof, Principal Investigator — Urology Department, Sheba Medical Center
Locations (1):
- Male Fertility Clinic, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Result] Ishijima SA, Okuno M, Mohri H. Zeta potential of human X- and Y-bearing sperm. Int J Androl. 1991 Oct;14(5):340-7. doi: 10.1111/j.1365-2605.1991.tb01102.x. PMID 1794918
- [Result] Chan PJ, Jacobson JD, Corselli JU, Patton WC. A simple zeta method for sperm selection based on membrane charge. Fertil Steril. 2006 Feb;85(2):481-6. doi: 10.1016/j.fertnstert.2005.07.1302. PMID 16595231